CLINICAL TRIAL: NCT03817489
Title: Starting From the Mind or the Body in Mind-Body Intervention: A Randomized Controlled Trial on Comparative Effectiveness of Mindfulness Meditation and Qigong on Psychophysiological Outcomes in Colorectal Cancer Patients
Brief Title: Mindfulness Meditation and Qigong for Colorectal Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17611615
Record Dates: First submitted 2019-01-10; First posted 2019-01-25 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer Survivors; Qigong; Mindfulness meditation; Randomized controlled trial; Cortisol
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: Baduanjin qigong (Experimental): This arm of participants will be receiving the Baduajin qigong intervention.
  Interventions: Behavioral: Baduanjin qigong
- Intervention: Mindfulness meditation (Experimental): This arm of participants will be receiving the Mindfulness meditation intervention.
  Interventions: Behavioral: Mindfulness meditation
- Control (No Intervention): This arm of participants will not receive any intervention and are allocated as a Wait-list Control group.

INTERVENTIONS:
Behavioral: Baduanjin qigong — The intervention consists of eight sequential forms of movements which is practiced with guidance on rhythmic breathing and mindful awareness. Each cycle of the eight movements requires 10 to 15 minutes for completion. Four cycles will be practiced in each session with short breaks arranged between them.
  Arms: Intervention: Baduanjin qigong
Behavioral: Mindfulness meditation — The intervention is developed based on the core components of the established Mindfulness-Based Stress Reduction and the Mindful Self-Compassion program with adaptation for local practice. The focus of the group is to nurture mindful awareness, acceptance, and self-compassion. The group sessions are composed of a combination of mindfulness-based practice, relaxation, and yoga exercise. The basic philosophy of this intervention is the emphasis of the nurturing of self-kindness attitude, and non-attachment attitude towards inter-personal connectedness and letting go of self-criticism, need for control, and defensive separation in times of adversity. Short breaks will be arranged between each practice.
  Arms: Intervention: Mindfulness meditation

SUMMARY:
Colorectal cancer imposes threats to patients' well-being. Although most physical symptoms can be managed by medication, psychosocial stressors may complicate survival and hamper quality of life. Mindfulness and Qigong, two kinds of mind-body exercise rooted in Eastern health philosophy, has been found effective in symptoms management, improving mental health, and reducing stress. With these potential benefits, a randomized controlled trial (RCT) is planned to investigate the comparative effectiveness of mindfulness and Baduanjin intervention on the bio-psychosocial wellbeing of people with colorectal cancer. A 3-arm RCT with waitlist control design will be used in this study. One hundred eighty-nine participants will be randomized into (i) Mindfulness, (ii) Baduanjin, or (iii) waitlist control groups. Participants in both the Baduanjin and mindfulness groups will receive 8-weeks of specific intervention. All three groups will undergo four assessment phases: (i) at baseline, (ii) at 4-week, (iii) at 8-week (post-intervention), and (iv) 6-month post-intervention (maintenance). All participants will be assessed in terms of cancer-related symptoms and symptom distress, mental health status, quality of life, stress level based on physiological marker. Based on prior research studies, participants in both the mindfulness and Baduanjn intervention group are expected to have better symptoms management, lower stress level, better mental health, and higher level of quality of life than the control group. This study contributes to better understanding on the common and unique effectiveness of mindfulness and Baduanjin qigong, as such patients and qualified healthcare professionals can select or provide practices which will produce maximum benefits, satisfaction, adherence, and sustainability.

DETAILED DESCRIPTION:
Colorectal cancer is one of the most common forms of cancer. Lifestyle modification and development of self-regulatory and self-care skills for maintaining psychological and physical well-being are especially important for recurrence prevention and long-term illness management. Mind-body practices are popular among cancer patients for being non-pharmacological, holistically beneficial, in addition to its feasibility for sustainable self-practice and self-care. Despite the popularity of practising qigong and mindfulness meditation among local patients, a systematic study on their effectiveness for cancer patients has yet to be conducted.

Qigong and mindfulness meditation represent two distinct forms of mind-body practices: dynamic and static. With both approaches attending to the breath, Qigong relies on physical exertion to arrive at mental and psychological changes while mindfulness meditation begins at mental level but can also impact physical health. Yet current knowledge on mind-body practices tells little about these contrasting approaches. Hence, this study not only aims to provide evidence for the psychophysiological effectiveness of qigong and mindfulness meditation for colorectal cancer patients, but also elucidate how these two fundamentally contrasting approaches differ in psychophysiological outcomes, rebalancing of dysfunctional cortisol rhythm, and affect long-term practice compliance.

Adopting a 3-arm randomized controlled trial design, this study will first independently study the effectiveness of Baduanjin qigong and Mindfulness meditation for Chinese colorectal cancer patients compared to controls on cancer-related symptoms and symptom distress, mental health, quality of life, biomarkers and mindfulness level. Another main objective is to examine the commonalities and differential effectiveness between a movement-based (Baduanjin qigong) and a mind-based (Mindfulness meditation) practice on the above outcomes, magnitude and pace of change, and the extended compliance throughout the 8-month study. A final objective is to examine the relationships among physical, psychological, and psychophysical variables and how these interactions between the mind and body. This study envisions advancing relationships change across the time.

189 Chinese-speaking patients with colorectal cancer will be recruited from local hospital and community organizations, then randomized into an 8-week (90-min/week) (i) Baduanjin qigong intervention, (ii) Mindfulness meditation intervention and (iii) No-intervention waitlist control. Participants will be assessed on 4 time points at (i) baseline prior randomization, (ii) mid-intervention (4th week), (iii) post-intervention (8th week) and (iv) 6 months post-intervention.

The measurement of both physiological and psychological outcomes will offer a comprehensive understanding on the mental and bodily changes after each intervention and their maintenance. Results will further support the reciprocal evidence-based mind-body practices which can be easily learned, self-practiced and incorporated into patients' lifestyles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary colorectal cancer of any stages 0 to III
* An expected survival length of 12 months or longer
* 0.5 to 5 years following completion of main treatment for colorectal cancer
* Ages 18 or higher
* Chinese speaking

Exclusion Criteria:

* Regularly practicing baduanjin qigong, other forms of qigong, taichi, meditation, mindfulness practices or yoga once a week or more
* Having participated in the above trainings in the past 6 months
* Severe cachexia, dizziness, bone pain, nausea or significant orthopedic problem or other contraindications for mild to moderate physical exertion
* Diagnosis of major medical or psychiatric disorder besides cancer (including but not limited to severe cardiovascular disease, epilepsy, uncontrolled diabetes, untreated hypothyroidism, delirium or dementia)
* Recurrence of colorectal cancer or other cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of Baseline Sleep Quality at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the Chinese version of Pittsburgh Sleep Quality Index (PSQI)
  * The PSQI is a self-report questionnaire that assesses multiple dimensions of seep over past one month.
  * The 19-item scale generates 7 'component' scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of the seven component scores yields one global score of subjective sleep.
Change of Baseline Cancer-related Symptom Distresses at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the the Chinese version of Memorial Symptom Assessment Scale (MSAS)
  * The scoring of the 32-item MSAS yields a MSAS Global Distress Index (10 items), the Physical Symptom Subscale score (12 items), the Psychological Symptom Subscale score (6 items), and a Total MSAS score.
Change of Baseline Health-related Quality of Life at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the Chinese (HK) version of the Short form-12 (SF-12)
  * This scale results in a physical and a mental health summary.
Change from Baseline Anxiety and Depressive symptoms at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the Cantonese/Chinese version of the Hospital Anxiety and Depression Scale (HADS)
  * The 14-item scale consists of two subscales (anxiety and depression) with seven items in each.
Change of Baseline Perceived stress at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the Chinese Perceived Stress Scale
  * This scale consists of 10 items about the degree to which life events are appraised as stressful.
Change of Baseline Mindfulness at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Administration of the Chinese Five Facet Mindfulness Questionnaire (Short form)
  * This scale has 5 domains, observing, describing, acting with awareness, nonjudging to inner experience and nonreacting to inner experience.
Change of Baseline Salivary cortisol level at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  * Salivary cortisol collection will be conducted by participants themselves.
  * Saliva samples will be collected at 5 prescribed times (awakening, 45 minutes post-awakening, 12:00pm, 5:00pm and 9:00pm) by placing a cotton swab under the tongue.
Change of Baseline Blood pressure at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  Measurement of both systolic and diastolic blood pressure.
Change of Baseline Heart rate at mid-intervention (week 4), post-intervention (week 8) and 6-month post-intervention | Baseline, Mid-Intervention (week 4), Post-intervention (week 8), 6-month Post-intervention
  Measurement of heart rate (beats per minute)
Change of Week 1 Practice Compliance at Week 2 to 7 of intervention, and 6-month post-intervention | Week 1 to Week 7 of intervention, and 6-month Post intervention
  Practice Compliance will be measured by participants' daily duration (minutes per week) of qigong or mindfulness meditation practice at Week 2, 3, 4, 5, 6 and 7 during the course of intervention group, and 6-month post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rainbow Tin Hung Ho, Principal Investigator — Department of Social Work and Social Administration, The University of Hong Kong
Locations (1):
- Centre on Behavioral Health, The University of Hong Kong, Hong Kong, Hong Kong

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03817489/Prot_SAP_000.pdf